CLINICAL TRIAL: NCT01435278
Title: Open-label Clinical Investigation to Evaluate the Safety and Efficacy of Glucosanol in Maintaining Body Weight Loss in Overweight and Obese Subjects
Brief Title: Efficacy and Safety of Glucosanol in Maintaining Body Weight
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INQ/017011
Record Dates: First submitted 2011-09-13; First posted 2011-09-16 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Overweight; Obesity
Keywords: Weight maintenance; BMI; Body weight; Overweight; Obesity; Satiety
MeSH Terms: conditions — Overweight; Obesity; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glucosanol (Active Comparator): 2 tablets 3 times a day
  Interventions: Device: Glucosanol

INTERVENTIONS:
Device: Glucosanol — 2 tablets taken 3 times a day.

SUMMARY:
To date, there is no clinical evidence on the efficacy and safety of Glucosanol in maintaining weight loss beyond the study duration of 12 weeks. The rationale for this open-label study is to assess the efficacy in preventing regain of loss body weight and safety of Glucosanol in subjects who are overweight or obese over a longer period after the initial weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled in, complied with, and completed the INQ/K/003411 (Glucosanol weight loss) study, with weight loss of at least 3% of baseline body weight
* Age 18 to 60 years at the time of inclusion into the INQ/K/003411 study
* BMI between 25-35 at the time of inclusion into the INQ/K/003411 study
* Expressed desire for weight maintenance
* Accustomed to 3 main meals per day
* Commitment to avoid the use of other weight loss products during study
* Females' agreement to use appropriate birth control methods during the active study period
* Subject declares in writing his/her consent to participate, understands requirements of the study and is willing to comply

Exclusion Criteria:

* Known sensitivity to the ingredients of the device (Phaseolus vulgaris or members of the Fabaceae family)
* History of diabetes mellitus • Fasting blood glucose more than 7 mmol/L
* History or clinical signs of endocrine disorders which may influence body weight (e.g. Cushing's disease, thyroid gland disorders)
* Clinically relevant excursions of safety parameter
* Current use of anti-depressants
* Presence of acute or chronic gastrointestinal disease (e.g. IBD, coeliac disease, pancreatitis)
* Uncontrolled hypertension (more than 160/110 mm Hg)
* Stenosis in the GI tract
* Bariatric surgery
* Abdominal surgery within the last 6 months prior to enrollment
* History of eating disorders like bulimia, anorexia nervosa within the past 12 months
* Other serious organ or systemic diseases such as cancer
* Any medication that could influence GI functions such as antibiotics, laxatives, opioids, glucocorticoids, anticholinergics, or anti-diarrheals
* Pregnancy or nursing
* Any medication or use of products for the treatment of obesity (e.g. Orlistat, other fatbinder, carb/starch blocker, fatburner, satiety products etc.)
* More than 3 hours strenuous sport activity per week
* History of abuse of drugs, alcohol or medication
* Smoking cessation within 6 months prior to enrolment
* Inability to comply due to language difficulties
* Presence of other factor(s) that, in the investigator's judgement, should preclude subject participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Body weight | 24 weeks
  Measured in kg using a calibrated scale

SECONDARY OUTCOMES:
Waist and hip circumference (cm) | 24 weeks
  Changes from baseline to end of study
Body mass index, BMI (kg/m2) | 24 weeks
  Changes from baseline to end of study
Body fat content and fat free mass | 24 weeks
  Changes from baseline to end of study
Effect on appetite, hunger and food cravings | 24 weeks
  The Control of Eating Questionnaire (COEQ) is used
Feeling of satiety | 24 weeks
  A 4-point categorical scale is used
Evaluation of the efficacy of Glucosanol by the subjects | 24 weeks
  A 4-point categorical scale is used
Full blood count | 24 weeks
  Done at baseline and end of study
Clinical chemistry parameter | 24 weeks
  Done at baseline and end of study
Blood pressure | 24 weeks
  Measured in mm Hg
Global evaluation of the safety of Glucosanol by the subjects | 24 weeks
  A 4-point categorical scale is used.
Global evaluation of the safety of Glucosanol by the investigators | 24 weeks
  A 4-point categorical scale is used
Occurrence of adverse events | 24 weeks
  All reported adverse events, regardless of causality, will be recorded in the source documents and case report forms

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Grube, MD, Berlin, Germany

REFERENCES:
- [Derived] Grube B, Chong WF, Chong PW, Riede L. Weight reduction and maintenance with IQP-PV-101: a 12-week randomized controlled study with a 24-week open label period. Obesity (Silver Spring). 2014 Mar;22(3):645-51. doi: 10.1002/oby.20577. Epub 2013 Sep 5. PMID 24006357